CLINICAL TRIAL: NCT00003237
Title: Phase II Trial of Post-Operative Adjuvant Paclitaxel + Cisplatin in Patients With Adenocarcinoma of the Esophagus, Gastro-Esophageal Junction or Cardia
Brief Title: Combination Chemotherapy After Surgery in Treating Patients With Cancer of the Esophagus or Stomach
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Group Chair, Eastern Cooperative Oncology Group
Purpose: Treatment
Other Study IDs: CDR0000066109; E-8296
Record Dates: First submitted 1999-11-01; First posted 2004-08-25 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Esophageal Cancer; Gastric Cancer
Keywords: stage II gastric cancer; stage III gastric cancer; stage II esophageal cancer; stage III esophageal cancer; adenocarcinoma of the stomach; adenocarcinoma of the esophagus
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Adenocarcinoma Of Esophagus | interventions — Cisplatin; Paclitaxel; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: cisplatin
Drug: paclitaxel
Procedure: surgical procedure

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug, and giving them after surgery, may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy, consisting of paclitaxel and cisplatin, given after surgery in treating patients with cancer of the esophagus or stomach.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the disease free survival and overall survival of patients with adenocarcinoma of the esophagus, gastroesophageal junction, or cardia receiving post-operative adjuvant paclitaxel plus cisplatin.

OUTLINE: Patients undergo esophagogastrectomies within 4-12 weeks prior to the study. Patients receive intravenous paclitaxel over 3 hours on day 1, followed by intravenous cisplatin. Treatment is repeated every 21 days for 4 courses. Patients exhibiting disease recurrence or unacceptable toxic effects are removed from the study. Patients are followed every 3 months for 2 years, every 6 months for the next 3 years, and then every 12 months thereafter.

PROJECTED ACCRUAL: A total of 55 patients will be accrued within 16 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven adenocarcinoma of the esophagus, gastroesophageal junction or cardia T2N1, T3 any N, T4 any N, and negative margins Proximal and distal margins of resection must be negative No metastases Must be within 4-12 weeks from date of surgery and clinically without evidence of local-regional or distant recurrence

PATIENT CHARACTERISTICS: Age: 18 and over Performance Status: ECOG 0-1 Life Expectancy: Not specified Hematopoietic: Absolute granulocyte count at least 1,500/mm3 Platelet count at least 120,000/mm3 Hepatic: SGOT no greater than 2 times upper limit of normal (ULN) Bilirubin no greater than 2 times ULN Renal: Creatinine within institutional normal limits Cardiovascular: No New York Heart Association class III or IV heart disease No symptomatic coronary artery disease No myocardial infarction within 6 months No clinically significant conduction system abnormalities such as second or third degree heart block or bundle branch block Neurologic: No symptomatic peripheral neuropathy No psychosis Other: Not pregnant or nursing Effective contraceptive method must be used by fertile patients No significant hearing loss No concurrent uncontrolled infection or medical illness No concurrent malignancies within 3 years, except: Nonmelanoma skin cancer Carcinoma in situ of the cervix No history of allergy to drugs containing cremophor No hypersensitivity to E. coli derived proteins

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent immunotherapy Chemotherapy: No prior chemotherapy No other concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy No concurrent radiotherapy Surgery: See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 1998-06-22 (Actual); Primary Completion 2003-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arlene A. Forastiere, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (30):
- United States (28):
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Lakeside), Chicago, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Central Illinois, Springfield, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Ochsner, New Orleans, Louisiana
  - New England Medical Center Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Veterans Affairs Medical Center - New York, New York, New York
  - Kaplan Cancer Center, New York, New York
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Ireland Cancer Center, Cleveland, Ohio
  - CCOP - St. Francis Hospital/Natalie Warren Bryant Cancer Center, Tulsa, Oklahoma
  - Allegheny University Hospitals- Hahnemann, Philadelphia, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - Veterans Affairs Medical Center - Madison, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin
- Veterans Affairs Medical Center - San Juan, San Juan, Puerto Rico
- Pretoria Academic Hospital, Pretoria, South Africa

REFERENCES:
- [Result] Armanios M, Xu R, Forastiere AA, Haller DG, Kugler JW, Benson AB 3rd; Eastern Cooperative Oncology Group. Adjuvant chemotherapy for resected adenocarcinoma of the esophagus, gastro-esophageal junction, and cardia: phase II trial (E8296) of the Eastern Cooperative Oncology Group. J Clin Oncol. 2004 Nov 15;22(22):4495-9. doi: 10.1200/JCO.2004.06.533. PMID 15542799